CLINICAL TRIAL: NCT03421964
Title: Intervention to Promote Survivor Resilience and Adjustment: Efficacy and Sustainability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20011840; 90DPTB0005 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience/Adjustment Counseling (Active Comparator): Intervention to promote resilience and adjustment (RAI) - The RAI was developed based upon considerable clinical experience and research review. The RAI is a structured approach to helping individuals after traumatic brain injury address issues related to resilience and adjustment to injury. The RAI is implemented in seven, 60-minute, virtual sessions.
  Interventions: Behavioral: Resilience/Adjustment Counseling
- Resilience/Adjustment Counseling with Booster Sessions (Experimental): Intervention to promote resilience and adjustment (RAI) is implemented in seven, 60-minute, virtual sessions; however individuals within this study arm will receive three additional 60-minute, virtual sessions three months after completing the seven initial sessions. The three booster sessions provide an opportunity for individuals to review course content, consolidate gains, and discuss challenges.
  Interventions: Behavioral: Resilience/Adjustment Counseling with Booster Sessions

INTERVENTIONS:
Behavioral: Resilience/Adjustment Counseling — The Resilience and Adjustment Intervention (RAI) consists of seven 60-minute sessions scheduled over seven weeks. Before the first session, participants will be mailed an empty loose-leaf binder to store and organize completed self-assessments, reading materials, and homework assignments from each session. They will be asked to review materials and complete worksheets between sessions. The RAI will be implemented by experienced, licensed therapists.
  Other Names: RAI
  Arms: Resilience/Adjustment Counseling
Behavioral: Resilience/Adjustment Counseling with Booster Sessions — The Resilience and Adjustment Intervention (RAI) consists of seven 60-minute sessions scheduled over seven weeks. Before the first session, participants will be mailed an empty loose-leaf binder to store and organize completed self-assessments, reading materials, and homework assignments from each session. They will be asked to review materials and complete worksheets between sessions.
  For the "RAI+" participants, three booster sessions will be implemented. The three weekly booster sessions will be scheduled to start three months following completion of Session 7 of the RAI. The program will be implemented by experienced, licensed therapists.
  Other Names: RAI+
  Arms: Resilience/Adjustment Counseling with Booster Sessions

SUMMARY:
The aims of this traumatic brain injury (TBI) study are:

1. to evaluate the short and long-term efficacy of two structured outpatient intervention programs, Resilience and Adjustment Intervention (RAI) vs. RAI with follow up booster sessions (RAI+) on resilience
2. to evaluate the short and long-term impact of intervention on emotional well-being and postinjury adjustment with the RAI vs. the RAI+
3. to evaluate the short and long-term impact of the RAI and the RAI+ on abilities including problem solving, communication, and stress management
4. to determine if demographic, lifestyle, injury, or treatment response information can predict maintenance of gains

DETAILED DESCRIPTION:
Participants will be assigned to either of two treatment groups: (1) Resilience and Adjustment Intervention (RAI), or (2) RAI+. After randomization, a second appointment will be scheduled. All participants will begin the 7-session treatment during their second appointment. The intervention consists of seven 60-minute sessions scheduled over seven weeks (see attached RAI Implementation Manual). The intervention will be implemented by experienced, licensed therapists (Ph.D. level Interventionists). Participants will be randomly assigned to one of the therapists.

The RAI and RAI+ groups will both complete the post-treatment measures immediately after the seventh treatment session and then 3, 4, and 9 months later. Data collection at 3, 4, and 9 months post-treatment will be completed via phone.

Furthermore, the RAI+ group will complete 3 booster sessions, spaced approximately 7-10 days apart, beginning 3 months after completion of the seventh treatment session (booster sessions will occur between the 3 and 4 month data collection described above).

Data will be analyzed to identify any therapist effects, as well as treatment effects. For the RAI and RAI+ groups, demographic, injury severity, and history information will be collected at intake using standard procedures and protocols. All participants will complete the 4 outcome measures (Connor-Davidson Resilience Scale, CD-RISC; Mayo Portland Adaptability Inventory-4, MPAI-4; 13 Item Stress Test; and Brief Symptom Inventory-18, BSI-18) at 5 time points (intake, post-treatment, and 3, 4 and 9 month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Mild, moderate, or severe TBI defined as: damage to brain tissue caused by an external mechanical force as evidenced by loss of consciousness due to brain trauma, post-traumatic amnesia (PTA), skull fracture, or objective neurological findings that can be reasonably attributed to TBI on physical examination or mental status examination.
* At least 3 months post-TBI.

Exclusion Criteria:

* Active substance abusers (e.g., intoxicated at arrival to intake).
* Individuals at imminent risk of psychiatric hospitalization, or in imminent danger of hurting themselves or others, as judged by the investigators, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy HSU, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Resilience/Adjustment Counseling With Booster Sessions: Intervention to promote resilience and adjustment (RAI) is implemented in seven, 60-minute, virtual sessions; however individuals within this study arm will receive three additional 60-minute, virtual sessions three months after completing the seven initial sessions. The three booster sessions provide an opportunity for individuals to review course content, consolidate gains, and discuss challenges.
  Resilience/Adjustment Counseling with Booster Sessions: The Resilience and Adjustment Intervention (RAI) consists of seven 60-minute sessions scheduled over seven weeks. Before the first session, participants will be mailed an empty loose-leaf binder to store and organize completed self-assessments, reading materials, and homework assignments from each session. They will be asked to review materials and complete worksheets between sessions.
  For the "RAI+" participants, three booster sessions will be implemented. The three weekly booster sessions will be scheduled to start three months following completion of Session 7 of the RAI. The program will be implemented by experienced, licensed therapists.
Period: Overall Study
Arm/Group | Resilience/Adjustment Counseling | Resilience/Adjustment Counseling With Booster Sessions
Started | 89 | 95
Completed | 66 | 69
Not Completed | 23 | 26
Not completed — Lost to Follow-up | 11 | 21
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Incarcerated | 1 | 0
Not completed — Inpt Treatment Facility | 1 | 1
Not completed — Virtual Platform Issues | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Resilience/Adjustment Counseling | Resilience/Adjustment Counseling With Booster Sessions | Total
Number analyzed (Participants) | 89 | 95 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.66) | 44.41 (13.39) | 44.36 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 44 | 97
  Male | 36 | 51 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 85 | 93 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 21 | 46
  White | 60 | 72 | 132
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 89 | 95 | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Completing the Two Structured Outpatient Intervention Programs Resilience and Adjustment Intervention (RAI) vs. RAI With Follow-up Booster Sessions (RAI+) on Resilience
Description: Evaluate the short and long-term efficacy of two structured outpatient intervention programs Resilience and Adjustment Intervention (RAI) vs. RAI with follow-up booster sessions (RAI+) on resilience. The RAI is implemented in a seven-session format with two or three topics covered during each 60-minute session. Sessions focus on skill-building to help clients enhance existing skills and develop new skills; psychological support through offering empathy, encouragement, and hope; and education via instruction and discussion. This measure is being quantitatively measured by the number of subjects that completed the assessment for each arm.
Time Frame: Data collection will be after the 7th treatment session and at 3,4 and 9 months post-treatment
Population: Number of participants who have completed the treatment sessions for each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Resilience/Adjustment Counseling | Resilience/Adjustment Counseling With Booster Sessions
Number analyzed (Participants) | 20 | 16
Participants | 12 | 0

2. Secondary Outcome: Mayo Portland Adaptability Inventory-4 (MPAI-4)
Description: Adjustment Subscale reflects emotional self-regulation; items relate to anxiety, depression, irritability, anger, social interaction, and self-awareness. Raw scores range from 0-46. Ability Subscale reflects cognitive and physical abilities, including verbal and nonverbal communication and problem-solving abilities. Raw scores range from 0-47. Adjustment Subscale: higher scores indicate greater severity. Ability Subscale: higher scores indicate greater problem severity. T scores between 40 and 60 would be considered average of people involved in rehabilitation following brain injury. T-scores between 40 and 50 may be considered in the mild to moderate range of overall severity compared to other people with ABI.; T-scores between 50 and 60, in the moderate to severe range. T-scores above 60 would suggest severe limitations even as compared to other people with ABI. T-scores between 30 and 40 suggest mild limitations. T-scores below 30 represent relatively good outcomes.
Time Frame: Change from Baseline to Follow-Up (11 months after Baseline)
Population: Subjects
Measure: Mean (Standard Deviation); unit: Change in BSI T-scores (mean=50, sd=10)
Arm/Group | Resilience/Adjustment Counseling | Resilience/Adjustment Counseling With Booster Sessions
Number analyzed (Participants) | 51 | 67
Change in BSI T-scores (mean=50, sd=10) | -3.07 (5.42) | -4.42 (6.00)

3. Secondary Outcome: Brief Symptom Inventory-18 (BSI-18), 18-item Self-report Instrument Was Developed to Quantify Psychological Distress in the General Population
Description: The BSI-18 is used because of its sound psychometric properties, and global assessment of psychological issues commonly found in individuals with TBI. Frequency ratings for items in three primary symptom dimensions (Somatization, Depression, and Anxiety) are added to yield the Global Severity Index (GSI). The GSI score reflects the overall distress level and is the focus of the present investigation. Frequency ratings for items in three primary symptom dimensions (Somatization, Depression, and Anxiety) are added to yield the Global Severity Index (GSI). T-scores are calculated based on community norms (50 indicates the population mean with a standard deviation of 10). Higher T scores are indicative of greater symptom severity. Somatization subscale: (Raw scores range from 0-19+), Depression subscale: (Raw scores range from 0-23+), Anxiety subscale: (Raw scores range from 0-20+), Global Severity Index: (Raw scores range from 0-53+)
Time Frame: Change from Baseline to Follow-Up (11 months after Baseline)
Measure: Mean (Standard Deviation); unit: Change in BSI T-scores (mean= 50; SD=10)
Arm/Group | Resilience/Adjustment Counseling | Resilience/Adjustment Counseling With Booster Sessions
Number analyzed (Participants) | 51 | 67
Change in BSI T-scores (mean= 50; SD=10) | -7.6 (8.62) | -7.72 (11.28)

4. Secondary Outcome: 13 Item Stress Test
Description: This self-report measure was developed more than a decade ago for clinical research studies on stress management with survivors and caregiving family members. Sample items include, "I have more to do than I can handle," "I'm pushing myself too hard," and "I can't stand living like this." Items are rated as True (+1) or False (0) with higher scores indicating higher stress levels. The measure has been shown to be sensitive to family intervention after TBI.63,64 The Total Score is the measure of interest in the present investigation. Total raw score ranges from 0-13. Higher raw scores are indicative of increased distress. There are no subscales used in this measure.
Time Frame: Change from Baseline to Follow-Up (11 months after Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resilience/Adjustment Counseling | Resilience/Adjustment Counseling With Booster Sessions
Number analyzed (Participants) | 49 | 63
units on a scale | -1.47 (2.36) | -1.9 (2.77)

ADVERSE EVENTS:
Time Frame: Through the intervention (seven weeks) and an additional 12 months for follow-up
Arm/Group | Resilience/Adjustment Counseling | Resilience/Adjustment Counseling With Booster Sessions
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/26
Other Adverse Events (participants affected / at risk) | 0/22 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT03421964/Prot_SAP_002.pdf
  • Informed Consent Form (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT03421964/ICF_003.pdf